CLINICAL TRIAL: NCT04871919
Title: A Prospective, Non-interventional Study of the Effectiveness, Safety, and Health Related Outcomes in Patients With Moderate to Severe Active Rheumatoid Arthritis Receiving Filgotinib
Brief Title: Prospective Observational Study of Filgotinib in Subjects With Rheumatoid Arthritis
Acronym: FILOSOPHY
Status: Active, not recruiting | Type: Observational
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: GLPG0634-CL-401; 48323 (Other: HMA-EMA Catalogues)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: filgotinib; safety; effectiveness; patient reported outcome
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Filgotinib: Individuals will receive treatment for moderate to severe active rheumatoid arthritis with at least one dose of filgotinib in accordance with the product label
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablets are administered in accordance with the product label
  Other Names: Jyseleca

SUMMARY:
An observational study to describe the effectiveness, safety, and patient-reported outcomes in patients with moderate to severe active rheumatoid arthritis (RA) receiving filgotinib in real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years with a diagnosis of moderate to severe active RA being prescribed filgotinib in accordance with the local standard of care and product label for the first time.
* Patients must be willing and able to use an electronic device to complete the study patient-reported outcome (PRO).

Exclusion Criteria:

- Participation in any other interventional or non-interventional study without prior approval from the Medical Monitor. This does not preclude inclusion of patients enrolled to national registries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients aged ≥ 18 years with moderate to severe active RA receiving filgotinib who will be enrolled across participating countries within Europe.
Sampling Method: Non-Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Treatment persistence rates | Up to 24 months
  To evaluate the treatment persistence rate at 24 months, defined as the rate of patients continuing to receive filgotinib 24 months from treatment initiation.

SECONDARY OUTCOMES:
patients' assessment of pain, Visual Analogue Scale (Pain VAS) | Up to 24 months; it will be evaluated as exploratory objectives in the optional 24-months extension period; i.e. at approximately 30, 36, 42, and 48 months.
patients' assessment of fatigue, Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F score) | Up to 24 months; it will be evaluated as exploratory objectives in the optional 24-months extension period; i.e. at approximately 30, 36, 42, and 48 months.
patients' assessment of Work Productivity and Activity Impairment: Rheumatoid Arthritis (WPAI-RA) | Up to 24 months; it will be evaluated as exploratory objectives in the optional 24-months extension period; i.e. at approximately 30, 36, 42, and 48 months.
medication adherence, compliance questionnaire rheumatology 19 (CQR19) | Up to 24 months; it will be evaluated as exploratory objectives in the optional 24-months extension period; i.e. at approximately 30, 36, 42, and 48 months.
medication adherence, compliance questionnaire rheumatology 5 (CQR5) | Up to 24 months; it will be evaluated as exploratory objectives in the optional 24-months extension period; i.e. at approximately 30, 36, 42, and 48 months.
Number of adverse events and serious adverse events | Up to 24 months; it will be evaluated as exploratory objectives in the optional 24-months extension period; i.e. at approximately 30, 36, 42, and 48 months.
patients' assessment of Rheumatoid Arthritis Impact of Disease (RAID) | Up to 24 months; it will be evaluated as exploratory objectives in the optional 24-months extension period; i.e. at approximately 30, 36, 42, and 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alfasigma Study Director, Study Director — Alfasigma S.p.A.
Locations (89):
- Belgium (15):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - Imelda VZW, Bonheiden
  - AZ Sint-Jan Brugge-Oostende, Bruges
  - Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi asbl, Charleroi
  - UZ Antwerpen, Edegem
  - Reumacentrum Genk, Genk
  - Reumaclinic Genk, Genk
  - AZ Maria Middelares, Ghent
  - Reuma Instituut, Hasselt
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - ZNA Jan Palfijn, Merksem
  - CHU UCL Namur asbl - Site Godinne, Yvoir
- Germany (30):
  - Rheumazentrum Kupka, Altenburg
  - Praxis für Rheumatologie - Amberg, Amberg
  - Rheumatology Center Prof. Neeck, Bad Doberan
  - Charité Campus Mitte, Klinik für Rheumatologie und Klinische Immunologie, Berlin
  - Rheumatologische Schwerpunktpraxis, Berlin
  - Rheumapraxis am Schlachtensee, Berlin
  - Rheumapraxis Mexikoplatz, Berlin
  - Klinik fur Innere Medizin - Rheumatologie - Kreiskrankenhaus Demmin, Demmin
  - Rheumatologisches MVZ Dresden, Dresden
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Praxis Dilltal, Ehringshausen
  - MVZ Ambulantes Rheumazentrum Erfurt, Erfurt
  - Universitätsmedizin Greifswald, Abteilung Innere Medizin A, Greifswald
  - Internistisch-Rheumatologische Arztpraxis, Halle
  - Rheumatologie im Struenseehaus, Hamburg
  - Praxis für Rheumatologie, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumapraxis, Leipzig
  - Praxis für Internistische Rheumatologie, Leipzig
  - Rheumatologische Facharztpraxis, Magdeburg
  - Rheumapraxis, Mansfeld
  - Praxis far Rheumatologie, Gastroenterologie und Innere Medizin, München
  - Rheumatologisches Praxiszentrum St. Bonifatius, München
  - Rheumapraxis, Neubrandenburg
  - Medizinischen Versorgungszentrums für Rheumatologie, Planegg
  - Rheumahaus - GbR, Potsdam
  - Rheumazentrum Ratingen, Ratingen
  - Rheumatologisch-immunologische Arztpraxis, Templin
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Klinikverbund St. Antonius und St. Josef GmbH, Wuppertal
- Italy (10):
  - A.O.U. Policlinico di Bari, Bari
  - ASST degli Spedali Civili di Brescia, Brescia
  - AOU Policlinico Vittorio Emanuele-PO San Marco, Catania
  - A.O.U. di Ferrara - Nuovo ospedale S.Anna, Ferrara
  - S.C. Reumatologia Asl3, Genova
  - ASST Gaetano Pini CTO, Milan
  - Azienda Osp. Univ. Luigi Vanvitelli, Napoli
  - Policlinico Umberto I Univ. Sapienza, Roma
  - Policlinico Gemelli, Roma
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona
- Netherlands (9):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - READE, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Reumazorg Zuid West, Goes
  - Elkerliek Ziekenhuis, Helmond
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Erasmus MC, Rotterdam
  - Hagaziekenhuis, The Hague
  - Sint Maartenskliniek, Ubbergen
- Spain (12):
  - Complexo Hospitalario Universitario, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Hospital de Mérida, Mérida
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitari Son Espases, Palma
  - Hospital Provincial de Pontevedra, Pontevedra
  - Hospital Universitario Hospiten Rambla de Tenerife, Santa Cruz de Tenerife
  - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- United Kingdom (13):
  - Aberdeen Royal Infirmary PPDS, Aberdeen
  - Royal Free NHS Foundation Trust, Barnet
  - University Hospital Coventry, Coventry
  - Doncaster Royal Infirmary, Doncaster
  - Ninewells Hospital - PPDS, Dundee
  - Western General Hospital Edinburgh - PPDS, Edinburgh
  - Royal Liverpool University Hospital, Liverpool
  - Guy's and St Thomas NHS Foundation Trust - Guy's Hospital, London
  - Kings College Hospital, London
  - Luton and Dunstable Hospital, Luton
  - Freeman Hospital, Newcastle
  - Royal Berkshire Hospital NHS Foundation Trust, Reading
  - York Teaching Hospitals NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No